CLINICAL TRIAL: NCT02651636
Title: Effects of Combined Therapy With Myo-inositol and Alpha-Lipoic Acid on Clinical, Endocrine and Metabolic Features in Women Affected by Polycystic Ovary Syndrome
Brief Title: Combined Therapy With Myo-inositol and Alpha-Lipoic Acid in PCOS Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Rosanna Apa, Professor, Catholic University of the Sacred Heart
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 000102014
Record Dates: First submitted 2015-11-27; First posted 2016-01-11 (Estimated); Last update posted 2016-01-11 (Estimated); Status verified 2016-01

CONDITIONS: Polycystic Ovary Syndrome; Menstrual Pattern; Hyperandrogenism; Metabolic Features
MeSH Terms: conditions — Polycystic Ovary Syndrome; Hyperandrogenism | interventions — Inositol; Thioctic Acid; Folic Acid

ARMS (1):
- Open label (Experimental): Therapy with alpha-lipoic acid (800 mg), myoinositol (2000 mg) and folic acid (400 mcg) daily for six months
  Interventions: Drug: myo-inositol,alpha-lipoic acid and folic acid

INTERVENTIONS:
Drug: myo-inositol,alpha-lipoic acid and folic acid

SUMMARY:
The aim of our study is to investigate the effects of a combined treatment of alpha-lipoic acid and myoinositol on clinical, endocrine and metabolic features of women affected by PCOS. The study Group included 40 patients treated with a combined therapy of alpha-lipoic acid (800 mg), myoinositol (2000 mg) and folic acid (400 mcg) daily for six months. The investigation includes menstrual pattern, hirsutism score, hormonal assays, oral glucose tolerance test, lipidic profile at baseline and after six months of treatment.

ELIGIBILITY:
Inclusion Criteria:

* women with PCOS in accordance with Rotterdam criteria

Exclusion Criteria:

* pregnancy
* past history of cardiovascular disease,
* diabetes mellitus (or impaired glucose tolerance as determined by a standard 75 g oral glucose tolerance test),
* hypertension,
* significant liver or renal impairment,
* other hormonal dysfunction (hypothalamic, pituitary, thyroidal or adrenal causes for the clinical signs),
* neoplasms,
* unstable mental illness.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2014-06; Primary Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Number of cycles in six months of therapy | 6 months

SECONDARY OUTCOMES:
Hirsutism | 6 months
  Ferriman Gallwey score
Hyperandrogenism | 6 months
  Testosterone, Androstenedione, free androgen index
Insulin response to oral glucose tolerance test | 6 months
Lipidic profile | 6 months
  Total cholesterol, LDL cholesterol, HDL cholesterol, triglyceride